CLINICAL TRIAL: NCT03082560
Title: Design and Validation of a New Assessment Tool for Lichen Planopilaris, the Boston Grade of Activity in Lichen Planopilaris (Boston GOAL)
Brief Title: Design and Validation of a New Assessment Tool for Lichen Planopilaris
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Maryanne Makredes Senna, Dermatologist, Massachusetts General Hospital
Other Study IDs: 2016P002620
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Lichen Planopilaris of Scalp; Lichen Plano-Pilaris; Lichen Planopilaris; Frontal Fibrosing Alopecia
MeSH Terms: conditions — Lichen Planus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Healthy adult patients with lichen planopilaris
  Interventions: Diagnostic Test: Boston Grade of Activity in Lichen Planopilaris

INTERVENTIONS:
Diagnostic Test: Boston Grade of Activity in Lichen Planopilaris — A clinical assessment tool to objectively and accurately measure activity and severity in lichen planopilaris over time.

SUMMARY:
The study's Primary Objective is to design and validate a grading system for objective and accurate assessment of lichen planopilaris.

Secondary Objectives:

* To assess change in symptoms such as pain and itch using a Numeric Rating Scale(NRS) scores and quality of life using the Dermatology Life Quality Index (DLQI) scores
* To correlate this grading system with patient skin biopsies evaluating disease activity on a microscopic level
* To correlate this grading system with digital global photography and trichoscopy

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects in general good health between the ages of 18 and 80 years old
2. Clinical and histologic diagnosis of lichen planopilaris
3. Subject is able to understand and sign informed consent
4. Subject is able to complete the study and comply with study procedures
5. Subject has no known allergy to non-toxic ink
6. Subjects should be managed by an Massachusetts General Hospital dermatologist for their lichen planopilaris for the duration of the study

Exclusion Criteria:

Eligible subjects will be excluded from participation if they meet any of the following criteria:

1. Presence of dermatoses that might interfere with LPP diagnosis and/or evaluation such as seborrheic dermatitis or psoriasis
2. Other selected concomitant causes of hair loss, including discoid lupus erythematosus, central centrifugal cicatricial alopecia (CCCA), telogen effluvium
3. Abnormal TSH laboratory value >1 standard deviation above normal within last year
4. Any significant medical condition that may prevent the patient from participating in the study according to the investigator's assessment
5. Any known allergy to non-toxic ink Related to Biopsy
6. History of poor wound healing or blood-clotting abnormality
7. History of keloid formation or hypertrophic scarring
8. Regular intake of high doses of aspirin or anti-coagulant medications
9. Hypersensitivity to local anesthetics
10. History of poorly controlled diabetes mellitus
11. Pregnant, nursing or planning a pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy adult subjects with lichen planopilaris
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Boston Grade of Activity in Lichen Planopilaris (Boston GOAL) | 6 months
  Design and validate a grading system for objective and accurate assessment of lichen planopilaris.

CONTACTS AND LOCATIONS:
Overall Officials: Maryanne Senna, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No